CLINICAL TRIAL: NCT06505005
Title: RESTORE (Relieving Pain and Improving Sleep: Evaluating Topical Pain Relief and Sleep Patches to Optimize Effectiveness)
Brief Title: Relieving Pain and Improving Sleep: Evaluating Topical Pain Relief and Sleep Patches
Acronym: RESTORE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: SuperPatch Limited LLC (Industry)
Collaborators: Clarity Science LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RESTORE-001
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pain, Back; Pain, Acute; Sleep Disorder; Sleep Disorders, Circadian Rhythm; Sleep; Sleep Deprivation; Insomnia
Keywords: musculoskeletal pain; sleep disorder; insomnia; back pain; acute pain; sleep
MeSH Terms: conditions — Back Pain; Acute Pain; Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Sleep Deprivation; Sleep Initiation and Maintenance Disorders; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled, crossover trial with functional measurements
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active/Treatment (Active Comparator): Data will be collected at Baseline prior to first use of active patch (FREEDOM or REM) and then 7 days, and then at 14 days after use with the active patch. Baseline and Follow-up functional measurements will also be taken at 7 and 14 days after baseline.
  Interventions: Device: Drug- free, non-invasive patch (FREEDOM or REM Patch) with haptic vibrotactile trigger technology (VTT) Other Names:
- Non-Active/Control (Sham Comparator): Data will be collected at Baseline prior to first use of sham patch and then 7 days, and then at 14 days after use with the sham patch. Baseline and Follow-up functional measurements will also be taken at 7 and 14 days after baseline. Control group subjects will be crossed over to crossover group after completion of control group study period.
  Interventions: Device: Sham Patch without haptic vibrotactile trigger technology (VTT)
- Crossover (Active Comparator): Data will be collected at Baseline prior to first use of active patch (FREEDOM or REM) and then 7 days, and then at 14 days after use with the active patch. Baseline and Follow-up functional measurements will also be taken at 7 and 14 days after baseline for all arms.
  Interventions: Device: Drug- free, non-invasive patch (FREEDOM or REM Patch) with haptic vibrotactile trigger technology (VTT) Other Names:; Device: Sham Patch without haptic vibrotactile trigger technology (VTT)

INTERVENTIONS:
Device: Drug- free, non-invasive patch (FREEDOM or REM Patch) with haptic vibrotactile trigger technology (VTT) Other Names: — Drug- free, non-invasive patch (FREEDOM or REM Patch) with haptic vibrotactile trigger technology (VTT)
  Other Names: Haptic Vibrotactile Trigger Technology; VTT
  Arms: Active/Treatment; Crossover
Device: Sham Patch without haptic vibrotactile trigger technology (VTT) — Sham Patch without haptic vibrotactile trigger technology (VTT)
  Other Names: Sham Comparator
  Arms: Crossover; Non-Active/Control

SUMMARY:
This minimal risk, randomized, double-blind, placebo controlled Institutional Review Board (IRB)-approved study with functional measurements, will evaluate pain relief and sleep improvement after use of a drug- free, non-invasive patch (FREEDOM or REM Patch; The Super Patch Company Inc.); using validated scales and functional measurement tools along with crossover and control groups within the same subject group not receiving an 'active' patch.

DETAILED DESCRIPTION:
Emerging technologies that use haptic (skin pressure) technology have been studied and have shown positive improvements in stress levels, balance, sleep, and pain. The FREEDOM and REM patch (SuperPatch Company, Toronto, Canada and Florida, USA) that also incorporates this technology has shown promise to improve relieve pain and improve sleep. This IRB-approved, Randomized Controlled Trial (RCT) will measure effectiveness of the pain and sleep patches through assessment of validated scales and functional measurements such as the Brief Pain Inventory (BPI), the Schober Test, the Bubble Inclinometer Measurement, and the Flexion Finger-Floor Measurement for the pain patch, and Pittsburgh Sleep Quality Index (PSQI), the Insomnia Severity Index (ISI), and a sleep wearable monitor for the Sleep patch.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-64
* Ability to provide Informed Consent
* Received a study patch (active or sham) from their treating clinician (randomized) for back, shoulder, and other musculoskeletal pain.
* Has been diagnosed with an acute, moderate pain condition
* Agrees to wear an adhesive study patch during the study period

Exclusion Criteria:

* Patients who are beneficiaries of a government-funded healthcare program
* Use of drugs of abuse (illicit or prescription)
* Have an implanted device, or wears, or adheres any electrical device to the body during the study, other than a hearing aid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Severity | 14 days
  Changes in Pain Severity Score based on Brief Pain Inventory (BPI) for those subjects in Pain Arm and receiving the active patch (FREEDOM) or Control Sham patch. (PAIN SEVERITY SCORE: 0-10 Scale). Decrease in Severity Score indicates a decrease in pain severity.
Changes in Pain Interference | 14 days
  Changes in Pain Interference Score based on Brief Pain Inventory (BPI) or those subjects in Pain Arm and receiving the active patch (FREEDOM) or Control Sham patch. (PAIN INTERFERENCE SCORE: 0-10 Scale). Decrease in Interference Score indicates a decrease in pain interference.
Changes in Range of Motion and Flexibility | 14 days
  Changes in Range of Motion and Flexibility based on subject and clinician reporting for those subjects in Pain Arm and receiving the active patch (FREEDOM) or Control Sham patch. Subjects will be evaluated with a Schober test measurement (cm).
Changes in Range of Motion and Flexibility | 14 days
  Changes in Range of Motion and Flexibility based on subject and clinician reporting for those subjects in Pain Arm and receiving the active patch (FREEDOM) or Control Sham patch. Subjects will be evaluated with a Goniometer measurement (degree of rotation/360 and cm).
Changes in Range of Motion and Flexibility | 14 days
  Changes in Range of Motion and Flexibility based on subject and clinician reporting for those subjects in Pain Arm and receiving the active patch (FREEDOM) or Control Sham patch. Subjects will be evaluated with a Bubble Inclinometer measurement (degree of rotation/360).
Changes in Sleep Duration | 14 days
  Changes in Sleep Duration based on Pittsburgh Quality Sleep Index (PSQI) for those subjects in Sleep Arm and receiving the active patch (REM) or Control Sham patch.
Changes in Sleep Duration | 14 days
  Changes in Sleep Duration based on a measurement from a wearable device) for those subjects in Sleep Arm and receiving the active patch (REM) or Control Sham patch.
Changes in Sleep Quality | 14 days
  Changes in Sleep Quality based on Pittsburgh Quality Sleep Index (PSQI) for those subjects in Sleep Arm and receiving the active patch (REM) or Control Sham patch.
Changes in Sleep Interference | 14 days
  Changes in Sleep Interference Score based on Insomnia Severity Index (ISI) or those subjects in Sleep Arm and receiving the active patch (REM) or Control Sham patch.

SECONDARY OUTCOMES:
Changes in Pain Medication Use | 14 days
  Changes in Number of Pain Medications Used based on subject and clinician reporting for those subjects in Pain Arm and receiving the active patch (FREEDOM) or Control Sham patch during study period.
Changes in Sleep Medication Use | 14 days
  Changes in Number of Sleep Medication Used based on subject and clinician reporting for those subjects in Sleep Arm and receiving the active patch (REM) or Control Sham patch during the study period.
Changes in Awakenings during sleep | 14 days
  Changes in awakenings Use based on subject and clinician reporting for those subjects in Sleep Arm and receiving the active patch (REM) or Control Sham patch.

OTHER OUTCOMES:
Any side effects reported by patients will be documented and assessed by clinician and PI | 14 days
  Evaluation of reported side effects during study period based on self-report by subject or reported by clinician investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Fason, DO, Principal Investigator — Stein Medical Center
Locations (1):
- Stein Medical, Tyrone, Georgia, United States

REFERENCES:
- [Derived] Fason J, Hurwitz P, Gudin J. Reducing Pain and Improving Mobility Using Haptic Patch Technology: Results of the RESTORE Study. Pain Ther. 2025 Dec;14(6):1797-1807. doi: 10.1007/s40122-025-00780-0. Epub 2025 Oct 8. PMID 41057672